CLINICAL TRIAL: NCT03953729
Title: Effectiveness of Pre-emptive Analgesia in Children With Molar-incisor Hypomineralization (MIH): Triple-blind Clinal Study, Randomized and Controlled by Placebo
Brief Title: Effectiveness of Pre-emptive Analgesia in Children With Molar-incisor Hypomineralization (MIH)
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Vicioni-Marques, F, Fernanda Vicioni Marques, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AnalgesiaMIH
Record Dates: First submitted 2019-04-25; First posted 2019-05-17 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1:Ibuprofeno (Experimental): The child and his / her guardian shall immediately upon arrival for informed about the participation in the research, being evaluated on the criteria of inclusion and exclusion described above. Soon after the signature by the responsible for the child of the Informed Consent Form (Appendix A), the drug shall be administered at the dosage established by Clark's formula, according to the weight of each child. It will then be evaluated the degree of anxiety of the child in front of the dental treatment using the scale "Children's Fear Survey Schedule-Dental Subscale" (Barberio, 2017). After 30 minutes of drug administration, treatment will start.
  Interventions: Drug: Ibuprofen
- Group 2: Placebo (Placebo Comparator): The child and his / her guardian shall immediately upon arrival for informed about the participation in the research, being evaluated on the criteria of inclusion and exclusion described above. Soon after the signature by the responsible for the child of the Informed Consent Form (Appendix A), the placebo shall be administered at the dosage established by Clark's formula, according to the weight of each child. It will then be evaluated the degree of anxiety of the child in front of the dental treatment using the scale "Children's Fear Survey Schedule-Dental Subscale" (Barberio, 2017). After 30 minutes of drug administration, treatment will start.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen — The child and his / her guardian shall immediately upon arrival for informed about the participation in the research, being evaluated on the criteria of inclusion and exclusion described above. Soon after the signature by the responsible for the child of the Informed Consent Form (Appendix A), the drug shall be administered at the dosage established by Clark's formula, according to the weight of each child. It will then be evaluated the degree of anxiety of the child in front of the dental treatment using the scale "Children's Fear Survey Schedule-Dental Subscale" (Barberio, 2017). After 30 minutes of drug administration, treatment will start.
  Arms: Group 1:Ibuprofeno
Drug: Placebo — The child and his / her guardian shall immediately upon arrival for informed about the participation in the research, being evaluated on the criteria of inclusion and exclusion described above. Soon after the signature by the responsible for the child of the Informed Consent Form (Appendix A), the placebo shall be administered at the dosage established by Clark's formula, according to the weight of each child. It will then be evaluated the degree of anxiety of the child in front of the dental treatment using the scale "Children's Fear Survey Schedule-Dental Subscale" (Barberio, 2017). After 30 minutes of drug administration, treatment will start.
  Arms: Group 2: Placebo

SUMMARY:
Pain is defined by IASP (International Association for the Study of Pain) as "an unpleasant sensory and emotional experience associated with the damage actual or potential tissue or described in terms that suggest such harm". Episodes of pain and discomfort experienced by children are one of the main factors for fear and anxiety in dentistry, especially those that present the condition of Molar-Incisive Hipomineralization, where we observed increased levels of anxiety in relation to the treatment. In order to improve the painful sensation that patients with Molar-Incisor Hipomineralization present as well as anxiety demonstrated by these patients in face of dental treatment, the objective of present study will be to evaluate the occurrence and degree of pain after procedures dentists with administration of pre-emptive analgesia or placebo, in children with Molar-Incisive Hipomineralization. Fifty patients will be selected in the Pediatric Dentistry courses of the FORP-USP undergraduate course, aged 6 to 12 years, of both sexes, who present at least 2 (two) upper and / or lower molars affected by Molar- Incisors that need some kind of restorative treatment, extraction or endodontic treatment. Also, these patients should present enamel and dentin fractures caused by MIH, atypical restoration and / or atypical caries, and that present pain above the moderate degree (6>), after stimulation with air/water jet for 5 seconds.

ELIGIBILITY:
Inclusion Criteria:

* present at least 2 (two) upper molars and/or lower affected by Molar-Incisor Hypomineralization
* restorative treatment
* extraction
* endodontic treatment
* pain above the moderate degree (6>)

Exclusion Criteria:

* patients with suspected of analgesics of any type or presence of acute pain in the last 24 hours before the procedure
* patient with history of hepatopathy
* bleeding hemorrhagic disorders
* hypersensitivity to components
* patients and family members who do not have a telephone or that the children will not under parental supervision in the first 24 hours after care.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-10-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Visual Pain Scale | 24 hours
  The child will indicate in the Wong Baker Face Scale what was the face associated with his/her pain. This scale consists of a visual observation by the child of several faces represented in drawing, ranging from 0 (no pain) to 10 (unbearable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Fabrício K de Carvalho, Professor, Study Director — University of Sao Paulo, School of Dentistry of Ribeirão Preto
Locations (1):
- School of Dentistry of Ribeirao Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No